CLINICAL TRIAL: NCT01928030
Title: Pilot Phase 1-2 Investigational Study to Assess the Efficacy and Safety of Recombinant Hyaluronidase (rHUPH20) in the Treatment of Secondary Lymphedema Resulting From Local Management of Malignancy
Brief Title: Recombinant Human Hyaluronidase in Treating Lymphedema in Patients With Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Pegram, Susy Yuan-Huey Hung Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-27871; NCI-2013-01624 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRS0032 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2016-12

CONDITIONS: Lymphedema; Malignant Neoplasm
MeSH Terms: conditions — Lymphedema; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- recombinant human hyaluronidase (Experimental): Phase 1. 450 units recombinant human hyaluronidase (rHuPH20) administered SC on days 1, 3, 5, and 7 Phase 2: 900 units recombinant human hyaluronidase (rHuPH20) administered SC on days 1 to 21
  Interventions: Biological: recombinant human hyaluronidase

INTERVENTIONS:
Biological: recombinant human hyaluronidase — Given SC
  Other Names: Chemophase; rHuPH20

SUMMARY:
This phase 1-2 trial studies the side effects and the best dose of recombinant human hyaluronidase and to see how well it works in treating lymphedema in patients with cancer. Recombinant human hyaluronidase (r-hu-hyaluronidase, rHuPH20) may reduce limb edema size in patients with lymphedema.

DETAILED DESCRIPTION:
This is a phase 1, dose-escalation study followed by a phase 2 study.

Phase 1: rHuPH20 subcutaneously (SC) on days 1, 3, 5, and 7

Phase 2: rHuPH20 SC on days 1 to 21

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 2
* Unilateral upper limb secondary lymphedema
* Must have the ability to understand and the willingness to sign a written informed consent document
* Must agree to blood serum assessment including, complete blood count (CBC) with differential; comprehensive metabolic panel and serum osmolality at every sanctioned evaluation; additionally physician may require cardiac evaluation with echocardiogram, electrocardiogram, brain natriuretic peptide or urinalysis if deemed appropriate
* Must consent to multi-bio-frequency impedance analysis (MFBIA); the details are to be covered in consent
* Willing to sign consent for skin biopsies and phlebotomy
* Women of child bearing potential must have a documented negative pregnancy test within 2 weeks prior to day 1 of treatment and agree to use a non-hormonal form of birth control during the duration of the trial therapy

Exclusion Criteria:

* Pregnant or actively breast-feeding
* Bilateral upper extremity edema
* Bilateral manipulation of axilla within the last 24 months
* Active infections
* Receiving concomitant treatment for upper extremity lymphedema, or who have received treatment within the last 14 days
* Known allergic or hypersensitivity reaction to rHUPH20 or any hyaluronidase extracts
* Receiving concomitant diuretics or dihydropyridine class of calcium channel blockers; if an alternative medication is available, patient can become eligible after 3 half-lives of drug discontinued and patient remains medically stable
* Grade 2 or greater hypo-albuminemia, serum sodium greater than 150meq/L, serum osmolality greater than 300mOsm/kg or blood urea nitrate/serum creatinine ratio greater than 25, within 7 days of screening
* Unable or unwilling to self/home administer subcutaneous experimental drug; study nurse or physician will train individuals on proper administration techniques
* Unwilling or incapable of maintaining a detailed log of number of injections, the date, time and site of administration
* Active malignancy; those undergoing active treatment for malignancy in the adjuvant setting are eligible; treatment can include chemotherapy, targeted therapy or anti-hormonal therapy
* At least 4 weeks removed from surgery or radiation in affected arm
* Primary lymphedema; if edema can be explained by systemic or congenital illnesses, that patient will not be eligible for this study
* Must not have any concurrent condition which in the investigator's opinion makes it inappropriate for the patient to participate in the trial or which would jeopardize compliance with the protocol
* Must not have received any investigational agents within 30 days prior to commencing study treatment
* Active thrombophlebitis
* Pulmonary edema, congestive heart failure or pulmonary embolus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pegram, Principal Investigator — Stanford University; Stanley Rockson, Principal Investigator — School of Medicine
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- 450 Units rHuPH20 (Days 1, 3, 5, and 7): Patients receive 450 units rHuPH20 SC on days 1, 3, 5, and 7
- 900 Units rHuPH20 (Days 1, 3, 5, and 7): Patients receive 900 units rHuPH20 SC on days 1, 3, 5, and 7
- MTD rHuPH20 (Days 1 to 21): Days 1 to 21 Patients receive the maximum tolerated dose (MTD) of rHuPH20 SC on days 1 to 21.
Period: Overall Study
Arm/Group | 450 Units rHuPH20 (Days 1, 3, 5, and 7) | 900 Units rHuPH20 (Days 1, 3, 5, and 7) | MTD rHuPH20 (Days 1 to 21)
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hyaluronidase, Recombinant Human: Patients receive recombinant human hyaluronidase 450 units or 900 units SC on days 1, 3, 5, and 7 (Phase 1) and then on days 1 to 21 (Phase 2) in the absence of disease progression or unacceptable toxicity.
Arm/Group | Hyaluronidase, Recombinant Human
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 56 [56 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Adverse Events
Description: Reported as any untoward medical occurrence or worsening of a pre-existing medical condition in a participant administered recombinant human hyaluronidase, and judged possibly, probably, or definitely related to treatment
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Groups:
- 450 Units Recombinant Human Hyaluronidase (rHuPH20): Participants receive 450 units recombinant human hyaluronidase (rHuPH20) subcutaneously (SC) on Days 1, 3, 5, and 7 (Phase 1) and then on Days 1 to 21 (Phase 2) in the absence of disease progression or unacceptable toxicity.
Arm/Group | 450 Units Recombinant Human Hyaluronidase (rHuPH20)
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Reduction in Forearm Volume
Description: Number of patients that achieve a clinically significant reduction in lymphedema, assessed as a 20% reduction in excess forearm volume
Time Frame: Up to 1 year
Population: No participants received 900 units rHuPH20, and the MTD was not determined, so no participants received rHuPH20 at the MTD.
Measure: Count of Participants; unit: Participants
Arm/Group | 450 Units rHuPH20 (Days 1, 3, 5, and 7) | 900 Units rHuPH20 (Days 1, 3, 5, and 7) | MTD rHuPH20 (Days 1 to 21)
Number analyzed (Participants) | 3 | 0 | 0
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Recombinant Human Hyaluronidase: Participants who received 450 units recombinant human hyaluronidase (rHuPH20) subcutaneously in Phase 1 were assessed in this outcome measure, treatment-related adverse events.
  Biomarker analysis and pharmacology study were performed during study.
  recombinant human hyaluronidase: Given subcutaneously
Arm/Group | Recombinant Human Hyaluronidase
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human Hyaluronidase (N=3)
Erythema (injection site reaction) (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No